CLINICAL TRIAL: NCT02213328
Title: CHAMPS: Choices For Adolescent Prevention Methods For South Africa. Pilot Study B: 'PlusPills'
Brief Title: Acceptability, Safety, and Use of Daily Truvada Pre-Exposure Prophylaxis in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHAMPS PrEP; 11931 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Truvada (Experimental): All participants will take Truvada, once daily by mouth for the first 12 weeks of the study. After Week 12 of the study, only participants who indicate a willingness to use Truvada PrEP and who do not have any medical reasons not to do so will continue to receive the Truvada tablets through Week 52.
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — Fixed-dose combination tablet containing 200 mg of FTC plus 300 mg of TDF, taken once daily by mouth.
  Other Names: emtricitabine/tenofovir disoproxil fumarate, FTC/TDF

SUMMARY:
Truvada (emtricitabine/tenofovir disoproxil fumarate, or FTC/TDF) is a type of antiretroviral (ARV) medicine that is commonly used to treat HIV. Truvada is also used as pre-exposure prophylaxis (PrEP) to prevent HIV infection in HIV-negative adults. The purpose of this study is to evaluate the acceptability, safety, and use of daily Truvada PrEP as part of a comprehensive HIV prevention package in healthy, HIV-uninfected adolescents 15 to 19 years of age.

DETAILED DESCRIPTION:
Truvada PrEP is an approach used to protect HIV-uninfected adults against possible infection with HIV. The approach involves taking Truvada every day to prevent HIV infection in case the person is exposed to HIV (for example, through sex with an HIV-infected person). The purpose of this study is to evaluate the acceptability, safety, and use of daily Truvada PrEP as part of a comprehensive HIV prevention package in healthy, HIV-uninfected adolescents 15 to 19 years old. In addition to Truvada PrEP, the HIV prevention package will include HIV testing, management of sexually transmitted infections (STIs), risk reduction counseling, access to condoms, post-exposure prophylaxis (PEP), and circumcision counseling and referral for male participants.

The study will enroll 150 healthy, HIV-uninfected adolescents 15 to 19 years of age. The study will last for 12 months (52 weeks) and involve scheduled clinic visits at study entry (Week 0) and Weeks 4, 8, 12, 24, 36, 48, and 52.

For the first 12 weeks of the study, all participants will be provided with a supply of Truvada tablets to take once daily as part of the comprehensive HIV prevention package. At Weeks 12, 24, 36, and 48, participants will be offered the following options: to continue with the full HIV prevention package plus Truvada PrEP, to stop Truvada PrEP and continue with rest of the HIV prevention package, or to re-start Truvada PrEP if previously stopped. After Week 12 of the study, Truvada tablets will be given only to those participants who decide to take PrEP and who do not have any medical reasons not to do so. Regardless whether they choose to use Truvada PrEP after Week 12, all study participants will be followed through Week 52 of the study.

All study visits will include blood collection, counseling before and after HIV testing, urine collection for pregnancy testing (female participants only), completion of a sexual risk behavior questionnaire, receipt of a supply of condoms, contraceptive counseling, a medical history review, and disclosure of available test results. Select study visits may include a physical exam, blood and urine collection, testing and treatment of STIs, adherence counseling, and an acceptability assessment. Between Months 11 and 12 of the study, some participants will be randomly selected to participate in focus groups to discuss their experiences while taking Truvada PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 to 19 years (inclusive) at screening, verified per study site standard operating procedures (SOPs)
* Able and willing to provide written informed consent/assent (age dependent) to be screened for and to take part in the study
* Have a guardian who is able and willing to provide written informed consent for his or her child to be screened for and to take part in the study
* Able and willing to provide adequate locator information, as defined in site standard operating procedures (SOPs)
* HIV-uninfected based on testing performed by study staff at screening and enrollment
* Sexually active, as defined as a minimum of one act of (penile vaginal) sexual intercourse in the last 12 months, per self-report
* (For female participants) Negative pregnancy test at screening and enrollment and, per participant report, does not intend to become pregnant in the next 12 months
* (For female participants) Using an effective method of contraception at enrollment, and intending to use an effective method for the study duration; effective methods include low dose oral, implant, or injectable hormonal methods.
* Does not report intention to relocate out of the study area during the course of the study
* Does not have job or other obligations that would require long absences from the area (for more than 4 weeks at a time)
* Willing to undergo all study-required procedures
* At screening and enrollment, agrees not to participate in other research studies involving drugs or medical devices for the next 12 months

Exclusion Criteria:

Participants who meet any of the following criteria, at baseline, are excluded from the study:

* As determined by the Site Investigator, any significant uncontrolled active or chronic disease process such as but not limited to diabetes, hypertension, and other diseases involving the cardiovascular, pulmonary, gastrointestinal, genitourinary, musculoskeletal, and central nervous systems
* Confirmed Grade 2 or greater hypophosphatemia
* Presence of serious psychiatric symptoms (e.g., active hallucinations)
* Visibly distraught at the time of consent (e.g., suicidal, homicidal, exhibiting violent behavior)
* Intoxicated or under the influence of alcohol or other drugs at the time of consent
* Acute or chronic hepatitis B infection (i.e., if hepatitis B surface antigen positive)
* Hepatitis B seronegative and refuses vaccination
* Renal dysfunction (creatinine clearance less than 75 ml/min); Use Cockroft-Gault equation as detailed in the protocol
* Urine dipstick for protein and glucose, excluding values of "1 +" or greater
* Any history of bone fractures not explained by trauma
* Any Grade 2 or greater toxicity on screening tests and assessments
* Concurrent participation in an HIV vaccine study or other investigational drug study
* Known allergy/sensitivity to the study drug or its components
* Use of disallowed medications (as detailed in the protocol)

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda-Gail Bekker, MBChB, PhD, Principal Investigator — Desmond Tutu HIV Centre
Locations (2):
- South Africa (2):
  - Desmond Tutu HIV Foundation Non-Network CRS, Cape Town
  - Perinatal HIV Non-network Research CRS, Soweto

REFERENCES:
- [Derived] Gill K, Johnson L, Dietrich J, Myer L, Marcus R, Wallace M, Pidwell T, Mendel E, Fynn L, Jones K, Wiesner L, Slack C, Strode A, Spiegel H, Hosek S, Rooney J, Gray G, Bekker LG. Acceptability, safety, and patterns of use of oral tenofovir disoproxil fumarate and emtricitabine for HIV pre-exposure prophylaxis in South African adolescents: an open-label single-arm phase 2 trial. Lancet Child Adolesc Health. 2020 Dec;4(12):875-883. doi: 10.1016/S2352-4642(20)30248-0. Epub 2020 Oct 24. PMID 33222803

RESULTS

PARTICIPANT FLOW:
Groups:
- Truvada: All participants will take Truvada, once daily by mouth for the first 12 weeks of the study. After Week 12 of the study, only participants who indicate a willingness to use Truvada PrEP and who do not have any medical reasons not to do so will continue to receive the Truvada tablets through Week 48.
  Truvada: Fixed-dose combination tablet containing 200 mg of FTC plus 300 mg of TDF, taken once daily by mouth.
Period: Overall Study
Arm/Group | Truvada
Started | 148
Completed | 120
Not Completed | 28
Not completed — Withdrawal by Subject | 10
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 16

BASELINE CHARACTERISTICS:
Population: All participants are adolescent male and female 15-19 years old
Arm/Group | Truvada
Number analyzed (Participants) | 148
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 18 [17 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 148
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 148
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 148

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Report Willingness to Use the Study Regimen, Take up PrEP, and Remain on PrEP as Part of a Comprehensive Prevention Package
Description: The percentage of participants who report willingness to use the study regimen, take up PrEP, and remain on PrEP as part of a comprehensive prevention package measured at different time points in the study
Time Frame: Measured through Week 48
Population: Enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Truvada
Number analyzed (Participants) | 148
Participants
  Percentage of partcipants who reported willingness to use the study regimen | 148
  Percentage of participants who took up PrEP | 148
  Percentage of participants who remained on PrEP at 12 weeks | 122
  Percentage of participants who remained on PrEP at 24 weeks | 87
  Percentage of participants who remained on PrEP at 36 weeks | 85
  Percentage of participants who remained on PrEP at week 48 | 85

2. Primary Outcome: Number of Participants With Acceptability as Per Questionnaire Administered at Week 48
Description: Acceptability was assessed by asking partcipants if they liked truvada, at the week 48 visit
Time Frame: Measured at Week 48
Population: Participants attending week 48 visit and completing acceptability questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Truvada
Number analyzed (Participants) | 117
Participants | 97

3. Primary Outcome: Number of Adolescents Who Continue to Use PrEP (as Indicated by Dried Blood Spot [DBS] Levels) After the Initial 3-month Period
Description: Number of adolescents who continued to use PrEP (as indicated by dried blood spot level) after the initial 3-month period as indicated by DBS at week 24/36/48
Time Frame: Measured through Week 48
Measure: Count of Participants; unit: Participants
Groups:
- Truvada: All participants will take Truvada, once daily by mouth for the first 12 weeks of the study. After Week 12 of the study, only participants who indicate a willingness to use Truvada PrEP and who do not have any medical reasons not to do so will continue to receive the Truvada tablets through Week 48
  Truvada: Fixed-dose combination tablet containing 200 mg of FTC plus 300 mg of TDF, taken once daily by mouth.
Arm/Group | Truvada
Number analyzed (Participants) | 148
Participants
  Participants with truvada in DBS at week 24 | 74
  Participants with truvada in DBS at week 36 | 31
  Participants with truvada in DBS at week 48 | 22

4. Primary Outcome: Number of Participants With Grades 2, 3, and 4 Clinical and Laboratory Adverse Events
Description: Assessment of Grades 2, 3, and 4 clinical and laboratory adverse events measured through week 48 using the DAIDS table for grading adult and paediatric adverse events, dated Dec 2004, (clarification Aug 2009). Expedited Adverse Event (EAE) reporting followed standard reporting requirements as defined in the DAIDS Manual for Expedited Reporting of Adverse Events version 2·0, March 2011.
Time Frame: Measured through Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Truvada
Number analyzed (Participants) | 148
Participants
  Grade 2 | 14
  Grade 3 | 4
  Grade 4 | 2

5. Primary Outcome: Number of Adolescents Enrolled and Retained in the Study
Description: Count of participants who had been enrolled in the study and successfully completed the study
Time Frame: Measured through Week 52
Population: 15-19 year old boys and girls
Measure: Count of Participants; unit: Participants
Arm/Group | Truvada
Number analyzed (Participants) | 148
Participants
  Number of participants enrolled | 148
  Number of participants completing the study | 120

6. Secondary Outcome: Number of Participants Who Used PrEP at Any Time Point During the Study, Measured With Drug Levels at M4/8/12/24/36
Description: Number of participants who used oral PrEP at any time during the study and had drug levels present at any time point
Time Frame: Measured through Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Truvada
Number analyzed (Participants) | 148
Participants | 141

7. Secondary Outcome: Proportion of Adolescents With Detectable Drug Levels Who Report Using PrEP
Description: Proportion of adolescents with detectable drug levels who report using PrEP at weeks 12,24,36,48
Time Frame: Measured though Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Truvada
Number analyzed (Participants) | 148
Participants
  total enrolled participants | 148
  week 12 | 107
  week 24 | 74
  week 36 | 31
  week 48 | 22

8. Secondary Outcome: Number of Participants Reporting Multiple Partners in the Preceding Year as Evidenced by Participant Responses to Interviewer Administered Questionnaires at Enrolment
Description: Participants reporting multiple partners during interviewer administered questionnaires
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Truvada
Number analyzed (Participants) | 148
Participants | 49

9. Secondary Outcome: Reported Consistent Condom Use as Evidenced by Participant Responses to Interviewer-administered Questionnaires Adminstered at the Enrolment Visit
Description: Reported consistent condom use as evidenced by participant responses to interviewer-administered questionnaires
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Truvada
Number analyzed (Participants) | 148
Participants | 100

10. Secondary Outcome: Reported Alcohol and Substance Use as Evidenced by Participant Responses to Interviewer-administered Questionnaires at the Enrolment Visit
Description: Reported substance use and alcohol use as evidenced by participant responses to interviewer-administered questionnaires
Time Frame: Baseline visit
Measure: Count of Participants; unit: Participants
Arm/Group | Truvada
Number analyzed (Participants) | 148
Participants
  No. of participants reporting alcohol use | 83
  No. of participants reporting drug use | 25

11. Secondary Outcome: Percentage of Study Participants Who Seroconverted During the Study, Measured Until Month 52
Description: Frequency of HIV infection as measured by seroconversion of study participants during the approximate 12 months of follow up. HIV rapid testing was done in parallel using Determine™ HIV-1/2 Ag/Ab Combo and Uni-Gold™ Recombigen® HIV-1/2. If the rapid HIV test was reactive, an HIV-1 RNA qualitative assay (Abbot) was performed. A positive test was confirmed with a second blood sample collected a week later.
Time Frame: Measured through Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Truvada
Number analyzed (Participants) | 148
Participants | 1

ADVERSE EVENTS:
Time Frame: Grades 2, 3, and 4 clinical and laboratory adverse events collected over 1 year.
Arm/Group | Truvada
All-Cause Mortality (participants affected / at risk) | 0/148
Serious Adverse Events (participants affected / at risk) | 4/148
Other Adverse Events (participants affected / at risk) | 15/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Truvada (N=148)
Haemothorax (Injury, poisoning and procedural complications) | 1 (1) — Haemothorax secondary to stab chest. Unrelated to study product.
Para suicide attempt (Injury, poisoning and procedural complications) | 1 (1) — Participant took an overdose of truvada after a fight with her mother
Cholecystitis (Hepatobiliary disorders) | 1 (1) — Secondary to gallstones
Incarcerated peri-umbilical hernia (Gastrointestinal disorders) | 1 (1) — Required emergency surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Truvada (N=148)
Headache (Nervous system disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Drug Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Weight Loss (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-12-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT02213328/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT02213328/SAP_001.pdf
  • Informed Consent Form (2015-07-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT02213328/ICF_002.pdf